CLINICAL TRIAL: NCT00546182
Title: Phase 4 Study of Simvastatin That Affects Insulin Sensitivity
Brief Title: Simvastatin Reduces Adiponectin Levels and Insulin Sensitivity
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Other Study IDs: GMC-200405
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Hypercholesterolemia
Keywords: Lipophilic statins; Insulin resistance; hypercholesterolemic patients
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We hypothesized simvastatin may reduce adiponectin levels and insulin sensitivity in overweight hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein cholesterol levels more than 100 and body mass index more than 23.0

Exclusion Criteria:

* Patients with overt liver disease
* Chronic renal failure
* Hypothyroidism, myopathy
* Uncontrolled diabetes
* Severe hypertension, stroke
* Acute coronary events
* Coronary revascularization within the preceding 3 months, or
* Alcohol abuse.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: overweight hypercholesterolemic patients
Dates: Start 2004-01

PRIMARY OUTCOMES:
simvastatin may reduce adiponectin levels and insulin sensitivity in overweight hypercholesterolemic patients

CONTACTS AND LOCATIONS:
Overall Officials: Kwang K Koh, MD,PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gil Medical Center, Gachon University, Incheon, South Korea

REFERENCES:
- [Result] Yada T, Nakata M, Shiraishi T, Kakei M. Inhibition by simvastatin, but not pravastatin, of glucose-induced cytosolic Ca2+ signalling and insulin secretion due to blockade of L-type Ca2+ channels in rat islet beta-cells. Br J Pharmacol. 1999 Mar;126(5):1205-13. doi: 10.1038/sj.bjp.0702397. PMID 10205010